CLINICAL TRIAL: NCT05380505
Title: Examining Influence of Social Media Ads on Black and White Adolescents' Food Choices
Brief Title: Influence of Social Media Ads on Food Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 20-01796-1; R01CA248441 (NIH)
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Food Choices

STUDY DESIGN:
Intervention Model Description: The intervention is exposure to Facebook food ads that are either race congruent or race incongruent, and that have varying numbers of likes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1: Race Congruent Ads (Experimental): Participants will complete a 15-minute survey in which they will be randomized to view and rate Facebook food ads associated with their condition. Then they will complete a food purchasing task in which they will shop in an online store that will display six food items and six beverages. Finally, they will answer demographic questions (e.g., self-reported height and weight) and view a debriefing summary that describes the full purpose of the study.
  Interventions: Behavioral: Racially Congruent Ads
- Condition 2: Race Incongruent Ads (Experimental): Participants will complete a 15-minute survey in which they will be randomized to view and rate Facebook food ads associated with their condition. Then they will complete a food purchasing task in which they will shop in an online store that will display six food items and six beverages. Finally, they will answer demographic questions (e.g., self-reported height and weight) and view a debriefing summary that describes the full purpose of the study.
  Interventions: Behavioral: Racially Incongruent Ads

INTERVENTIONS:
Behavioral: Racially Congruent Ads — Facebook food ads that are racially congruent.
  Arms: Condition 1: Race Congruent Ads
Behavioral: Racially Incongruent Ads — Facebook food ads that are racially incongruent.
  Arms: Condition 2: Race Incongruent Ads

SUMMARY:
This is a randomized trial to examine the influence of race-congruent food marketing on social media among Black and White adolescents.

DETAILED DESCRIPTION:
This randomized trial evaluates the extent to which exposure to racially congruent vs. incongruent Facebook food ads causes Black vs. White adolescents to purchase more calories for a snack

ELIGIBILITY:
Inclusion Criteria:

* adolescent (13-17 years of age)
* who identifies as only non-Latino White or only Black/African American
* who logs into Facebook once daily
* who can read and speak English

Exclusion Criteria:

* participants who do not meet all criteria described above.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1252 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bragg, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads
Started | 588 | 550
Completed | 588 | 550
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads | Total
Number analyzed (Participants) | 588 | 550 | 1138
Age, Continuous [Mean (Full Range); unit: years] | 15 [13 to 17] | 15 [13 to 17] | 15 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 273 | 555
  Male | 306 | 277 | 583
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 47 | 106
  Not Hispanic or Latino | 529 | 502 | 1031
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 266 | 270 | 536
  White | 290 | 268 | 558
  More than one race | 27 | 10 | 37
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 588 | 550 | 1138

OUTCOME MEASURES:

1. Primary Outcome: Number of Calories Purchased
Time Frame: 15 minutes
Measure: Mean (Full Range); unit: calories
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads
Number analyzed (Participants) | 588 | 550
calories | 458 [117 to 750] | 477 [117 to 750]

2. Secondary Outcome: Attitude Toward Ad
Description: Attitude will be reported on a Likert scale of 1 to 100 (1 = likeable, 100 = unlikeable). The higher the score, the less likeable the ad is to the participant.
Time Frame: 15 minutes
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads
Number analyzed (Participants) | 588 | 550
score on a scale | 73.4 [0 to 100] | 68.7 [0 to 100]

3. Secondary Outcome: Time Spent Viewing Ad
Description: Time spend viewing ad.
Time Frame: 15 minutes
Measure: Mean (Full Range); unit: seconds
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads
Number analyzed (Participants) | 588 | 550
seconds | 10.3 [0.2 to 755.2] | 9.3 [0.1 to 236.9]

ADVERSE EVENTS:
Time Frame: 1 month
Description: non-systemic assessment
Arm/Group | Condition 1: Race Congruent Ads | Condition 2: Race Incongruent Ads
All-Cause Mortality (participants affected / at risk) | 0/588 | 0/550
Serious Adverse Events (participants affected / at risk) | 0/588 | 0/550
Other Adverse Events (participants affected / at risk) | 0/588 | 0/550

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT05380505/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT05380505/ICF_000.pdf